CLINICAL TRIAL: NCT06978985
Title: Adult SMA REACH: Development and Implementation of a Standardised Data Set and Data Collection Research Study in the UK Adult SMA Population
Brief Title: Adult SMA Research and Clinical Hub
Acronym: REACH
Status: Recruiting | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Newcastle University (Other); John Walton Muscular Dystrophy Research Centre (Unknown); Biogen (Industry); Roche Products Limited (Unknown)
Responsible Party: Principal Investigator, Chiara Marini Bettolo, Consultant Neurologist and Clinical Lead, Newcastle-upon-Tyne Hospitals NHS Trust
Other Study IDs: 9832
Record Dates: First submitted 2025-04-07; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Spinal Muscular Atrophy (SMA)
Keywords: SMA; Data collection; Adult SMA; SMA REACH; Data collection study; Spinal; Muscular Atrophy, Spinal; real-world data
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam; nusinersen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Spinal Muscular Atrophy: Participants over 16 years old with a genetically confirmed diagnosis of 5q SMA.
  Interventions: Drug: Risdiplam; Drug: Nusinersen Injectable Product

INTERVENTIONS:
Drug: Risdiplam — Risdiplam
  Other Names: Evrysdi
Drug: Nusinersen Injectable Product — Nusinersen
  Other Names: Spinraza

SUMMARY:
Adult SMA REACH is a data collection study aiming to gain a better understanding of the impact of standards of care and new treatments on the natural history of Spinal Muscular Atrophy (SMA). This study is sponsored by The Newcastle upon Tyne Hospitals NHS Foundation Trust. Adult SMA REACH is funded by Biogen and Roche.

Currently, there are three drug treatments available for SMA in the UK: Zolgensma, Nusinersen and Risdiplam. Zolgensma is the only approved drug - Nusinersen and Risdiplam are currently available as part of Managed Access Agreements (MAA).

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a genetic motor neuron disease with a broad spectrum of severity, affecting both infants and adults. Advances in treatment, including Nusinersen (Spinraza), onasemnogene abeparvovec (Zolgensma), and Risdiplam (Evrysdi), have significantly improved patient outcomes, highlighting the need for stronger clinical networks to monitor the long-term effects of these therapies.

The Adult SMA REACH Study builds upon the success of SMA REACH UK, which has been instrumental in collecting natural history and treatment data for paediatric SMA patients. The study benefits from collaboration with TREAT-NMD, the UK SMA Patient Registry, and iSMAC, aligning with international efforts to harmonise SMA data collection. By leveraging Newcastle University's experience in global SMA initiatives, Adult SMA REACH aims to enhance patient care, inform clinical decision-making, and contribute to future SMA research.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16 years (when patients will begin the transition process to adulthood)
* Genetically confirmed diagnosis of 5q SMA
* Signed informed consent to take part in the study

Exclusion Criteria:

* Non-5q SMA
* No genetic confirmation
* <16 years of age
* No signed informed consent or consent withdrawn

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with SMA will volunteer to participate in this study. The study will be advertised through neuromuscular disease clinics, the registry website, patient organisations and conferences throughout the UK and Ireland.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
World Health Organization (WHO) Motor Milestones | Baseline (at treatment initiation) and 6 monthly through study completion
  The WHO motor milestone assessment is a six-item checklist that dichotomously assesses whether a child can sit independently, crawl, stand with/without support, and walk with/without support. It is used in the Adult SMA population and in this study to categorise individuals as 'non-sitters', 'sitters' or 'walkers'. Changes in this score (loss or gain in function) and maintenance of score from baseline throughout treatment duration is assessed.
Revised Upper Limb Module (RULM) | Baseline (at treatment initiation) and 6 monthly through study completion
  The RULM is designed to capture upper limb function and consists of 19 items, and is scored out of 37 points (higher scores indicating better function).
6 Minute Walk Test (6MWT) | Baseline (at treatment initiation) and 6 monthly through study completion
  The 6MWT, which measures the distance a patient is able to walk within 6 min is used for only ambulant adult SMA patients in this study.
The Hammersmith Functional Motor Scale Expanded (HFMSE) | Baseline (at treatment initiation) and 6 monthly through study completion
  The HFMSE consists of 33 items, with a maximum of 66 points (higher scores indicating better function).
The Egen classification 2 (EK2) scale | Baseline (at treatment initiation) and 6 monthly through study completion
  The EK2 is a functional scale that includes 17 items for eight daily-life categories (wheelchair use, wheelchair transfers, trunk mobility, eating, swallowing, breathing, coughing, fatigue). Each item is scored from 0 to 3 for a maximum of 51 points (higher scores indicating worse function).

CONTACTS AND LOCATIONS:
Overall Officials: Prof Chiara Marini-Bettolo, MD, PhD, Principal Investigator — Newcastle-upon-Tyne Hospitals NHS Trust
Locations (18):
- United Kingdom (18):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - North Bristol NHS Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff and Vale University Health Board, Cardiff
  - NHS Greater Glasgow and Clyde, Glasgow
  - Bradford Teaching Hospitals NHS Foundation Trust, Leeds
  - The Walton Centre NHS Foundation Trust, Liverpool
  - University College London Hospitals NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - St George's University NHS Foundation Trust, London
  - Newcastle-upon-Tyne Hospitals NHS Trust, Newcastle upon Tyne
  - Nottingham University Hospitals Trust, Nottingham
  - The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry
  - Oxford University Hospitals Trust, Oxford
  - The Northern Care Alliance NHS Foundation Trust, Salford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - South West Wales Neuromuscular Service in Swansea, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://adultsmareach.co.uk/